CLINICAL TRIAL: NCT00272779
Title: A 96 Week Study Comparing the Antiviral Efficacy and Safety of Atazanavir/Ritonavir With Lopinavir/Ritonavir, Each in Combination With Fixed Dose Tenofovir-Emtricitabine in HIV-1 Infected Treatment in Naive Subjects
Brief Title: BMS-Reyataz Study in Treatment in Naive Subjects to Compare the Efficacy and Safety Between Boosted Reyataz and Kaletra When in Combination With Fixed Dose Truvada
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-138
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atazanavir (ATV) + Ritonovir (RTV) (Active Comparator): Participants were administered an oral dose of ATV 300 mg and RTV 100 mg once daily along with food on a background of fixed dose combination TDF 300 mg plus FTC 200 mg (TDF/FTC) once daily. Doses of ATV and RTV were taken 24 hours apart at the same time as the background TDF/FTC, up to 96 Weeks.
  Interventions: Drug: ATV; Drug: RTV; Drug: Tenofovi-Emtricitabine (TDF/FTC) tablet
- Lopinavir (LPV) + RTV (Active Comparator): Participants were administered an oral dose of LPV 400 mg and RTV 100 mg once daily along with food on a background of fixed dose combination TDF 300 mg plus FTC 200 mg (TDF/FTC) once daily. Doses of LPV and RTV were taken 24 hours apart at the same time as the background TDF/FTC, up to 96 Weeks.
  Interventions: Drug: RTV; Drug: Tenofovi-Emtricitabine (TDF/FTC) tablet; Drug: LPV

INTERVENTIONS:
Drug: ATV — 300mg Oral capsules for 96 weeks
  Other Names: Atazanavir; Reyataz; BMS-232632
  Arms: Atazanavir (ATV) + Ritonovir (RTV)
Drug: RTV — 100mg Oral Capsules for 96 weeks
Drug: Tenofovi-Emtricitabine (TDF/FTC) tablet — One tablet with 300 mg - 200 mg once a day for 96 weeks.
Drug: LPV — 400 mg (3 133mg capsules) BID for 96 weeks
  Arms: Lopinavir (LPV) + RTV

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and antiviral effects of atazanavir (ATV) plus ritonavir (RTV) versus a combination drug of lopinavir (LPV) plus RTV. A combination drug containing tenofovir (TDF) and emtricitabine (FTC) will also be taken by participants in both arms.

ELIGIBILITY:
Inclusion Criteria:

* HIV RNA ≥5000 c/ml

Exclusion Criteria:

* Any antiretroviral therapy within 30 days prior to screening;
* Women of Childbearing potential (WOCBP) unwilling or unable to use an acceptable method to avoid pregnancy for the entire study and for up to 8 weeks after the study;
* WOCBP using a prohibited contraceptive method
* WOCBP who are pregnant or breastfeeding;
* Women with a positive pregnancy test on enrollment or prior to study drug administration;
* Presence of a newly diagnosed HIV-Related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment;
* Suspected primary (acute) HIV infection;
* Prior antiviral therapy (>30 days of NRTI and/or >7 days of non-nucleoside reverse transcriptase inhibitor (NNRTI) or PI therapies) or any antiretroviral therapy within 30 days prior to screening; some exceptions are allowed for ARV therapy in use for Mother-to-child transmission;
* Participants with Cushing's syndrome;
* Untreated hypothyroidism or hyperthyroidism. A participant who is euthyroid on a stable replacement dose of thyroid hormone is acceptable provided the thyroid stimulating hormone (TSH) performed within 30 days of screening is within normal drug range;
* Recent therapy with agents with significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic or cytotoxic potential within 3 months of study start or expected need for such therapy at the time of enrollment; or therapy with methadone or ribavirin/interferons or treatment with neurotoxic drugs or drugs that affect CYP3A4;
* Participants with obstructive liver disease;
* Active alcohol or substance use sufficient, in the Investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis or chemical hepatitis;
* Proven or suspected acute hepatitis in the 30 days prior to study entry;
* Intractable diarrhea (≥6 loose stools/day for at least 7 consecutive days) within 30 days prior to study entry;
* Inability to swallow capsules;
* Active peripheral neuropathy;
* Presence of cardiomyopathy (due to any cause) or any significant cardiovascular disease, such as unstable ischemic heart disease;
* Known, clinically significant cardiac conduction system disease.
* Baseline laboratory values measured within 2 weeks prior to initiating study drugs as follows:

  1. calculated creatine clearance <60 mL/min as estimated by the Cockcroft-Gault equation;
  2. total serum lipase ≥ 1.4 times the upper limit of normal;
  3. liver enzymes (AST, ALT) ≥ 5 times the upper limit of normal;
  4. total serum bilirubin ≥ 1.5 times the upper limit of normal.
* Hypersensitivity to any component of the formulation of study drug;
* Prohibited therapies;
* Any other clinical conditions or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for study or unable to comply with the dosing requirements;
* Prisoners or participants who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- United States (8):
  - Local Institution, Phoenix, Arizona
  - Local Institution, Laguna Beach, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Dallas, Texas
  - Local Institution, Fort Worth, Texas
- Argentina (5):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
  - Local Institution, Córdoba
- Australia (3):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Carlton, Victoria
  - Local Institution, South Yarra, Victoria
- Local Institution, Vienna, Austria
- Belgium (2):
  - Local Institution, Bruges
  - Local Institution, Ghent
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Recife, Pernambuco
  - Local Institution, Campinas, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (2):
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Chile (2):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
- Local Institution, Bogotá, Colombia
- Local Institution, San José, Costa Rica
- Local Institution, Santo Domingo, Dominican Republic
- France (3):
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Villejuif
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Cologne
  - Local Institution, Hamburg
- Local Institution, Guatemala City, Guatemala
- Local Institution, Kowloon, Hong Kong
- Local Institution, Jakarta, Indonesia
- Italy (4):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Roma
  - Local Institution, Torino
- Mexico (7):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopal, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Chihuaha
  - Local Institution, Durango
  - Local Institution, San Luis Potisi
- Netherlands (2):
  - Local Institution, Maastricht
  - Local Institution, Utrecht
- Local Institution, Panama City, Panama
- Local Institution, Lima, Peru
- Local Institution, Lisbon, Portugal
- Puerto Rico (2):
  - Local Institution, Ponce
  - Local Institution, San Juan
- Local Institution, Singapore, Singapore
- South Africa (9):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Meadowdale, Gauteng
  - Local Institution, Westdene, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Mowbray, Western Cape
  - Local Institution, Parow, Western Cape
  - Local Institution, Rugby, Western Cape
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Córdoba
  - Local Institution, Madrid
  - Local Institution, Málaga
- Taiwan (2):
  - Local Institution, Kaohsiung City
  - Local Institution, Taipei
- Thailand (2):
  - Local Institution, Chiang Mai
  - Local Institution, Khonkaen
- United Kingdom (2):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester

REFERENCES:
- [Background] Molina JM, Andrade-Villanueva J, Echevarria J, Chetchotisakd P, Corral J, David N, Moyle G, Mancini M, Percival L, Yang R, Wirtz V, Lataillade M, Absalon J, McGrath D; CASTLE Study Team. Once-daily atazanavir/ritonavir compared with twice-daily lopinavir/ritonavir, each in combination with tenofovir and emtricitabine, for management of antiretroviral-naive HIV-1-infected patients: 96-week efficacy and safety results of the CASTLE study. J Acquir Immune Defic Syndr. 2010 Mar;53(3):323-32. doi: 10.1097/QAI.0b013e3181c990bf. PMID 20032785
- [Background] Molina JM, Andrade-Villanueva J, Echevarria J, Chetchotisakd P, Corral J, David N, Moyle G, Mancini M, Percival L, Yang R, Thiry A, McGrath D; CASTLE Study Team. Once-daily atazanavir/ritonavir versus twice-daily lopinavir/ritonavir, each in combination with tenofovir and emtricitabine, for management of antiretroviral-naive HIV-1-infected patients: 48 week efficacy and safety results of the CASTLE study. Lancet. 2008 Aug 23;372(9639):646-55. doi: 10.1016/S0140-6736(08)61081-8. PMID 18722869
- [Derived] Zhu L, Liao S, Child M, Zhang J, Persson A, Sevinsky H, Eley T, Xu X, Krystal M, Farajallah A, McGrath D, Molina JM, Bertz R. Pharmacokinetics and inhibitory quotient of atazanavir/ritonavir versus lopinavir/ritonavir in HIV-infected, treatment-naive patients who participated in the CASTLE Study. J Antimicrob Chemother. 2012 Feb;67(2):465-8. doi: 10.1093/jac/dkr490. Epub 2011 Nov 25. PMID 22121190
- [Derived] Uy J, Yang R, Wirtz V, Sheppard L, Farajallah A, McGrath D. Treatment of advanced HIV disease in antiretroviral-naive HIV-1-infected patients receiving once-daily atazanavir/ritonavir or twice-daily lopinavir/ritonavir, each in combination with tenofovir disoproxil fumarate and emtricitabine. AIDS Care. 2011 Nov;23(11):1500-4. doi: 10.1080/09540121.2011.565033. Epub 2011 Jul 7. PMID 21732894
- [Derived] Squires KE, Johnson M, Yang R, Uy J, Sheppard L, Absalon J, McGrath D. Comparative gender analysis of the efficacy and safety of atazanavir/ritonavir and lopinavir/ritonavir at 96 weeks in the CASTLE study. J Antimicrob Chemother. 2011 Feb;66(2):363-70. doi: 10.1093/jac/dkq457. Epub 2010 Dec 9. PMID 21148235

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1057 HIV-infected participants, 174 participants were not randomized to receive study drug, the main reason being that they did not meet the study criteria (133/174; 76%). 441 randomized to ATV received any drug and 437 randomized to LPV received any drug. 438 and 440 participants randomized to ATV and LPV, respectively, received correct drug.
Groups:
- ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD: Participants were administered an oral dose of Atazanavir (ATV) 300 mg and ritonavir (RTV) 100 mg once daily along with food. Doses were taken 24 hours apart at the same time as fixed dose combination tenofovir (TDF) 300 mg plus emtricitabine (FTC) 200 mg once daily.
- LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD: Participants were administered lopinavir (LPV) 400 mg or ritonavir (RTV) 100 mg twice daily along with food. Doses were taken approximately 12 hours apart while tenofovir (TDF) 300 mg once daily and emtricitabine (FTC) 200 mg once daily was administered at the same time as 1 of the 2 daily doses of LPV/RTV.
Period: Baseline Through Week 48
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Started | 440 (Number of participants randomized to ATV) | 443 (Number of participants randomized to LPV)
RECEIVED ANY TREATMENT | 441 (1 participant randomized to LPV received ATV instead (treatment error)) | 437 (3 participants received ATV instead of LPV (treatment error), 3 participants never treated with LPV)
TREATED AS RANDOMIZED | 438 | 440
Discontinued Before Week 48 | 39 | 58
Discontinued on or After Week 48 | 14 | 14
STILL ON TREATMENT | 385 | 368
Completed | 0 | 0
Not Completed | 440 | 443
Not completed — Adverse event before Week 48 | 10 | 14
Not completed — Death before Week 48 | 4 | 4
Not completed — Lack of efficacy before Week 48 | 5 | 8
Not completed — Lost to follow-up before Week 48 | 6 | 6
Not completed — Viral load rebound before Week 48 | 1 | 0
Not completed — Poor/non compliance before Week 48 | 6 | 9
Not completed — Pregnancy before Week 48 | 2 | 2
Not completed — No longer meets criteria before Week 48 | 1 | 0
Not completed — Withdrew consent before Week 48 | 4 | 13
Not completed — Participant's decision before wk 48 | 0 | 1
Not completed — Chose different site before wk 48 | 0 | 1
Not completed — Adverse event on/after Week 48 | 1 | 1
Not completed — Death on/after Week 48 | 1 | 1
Not completed — Lack of efficacy on/after Week 48 | 7 | 1
Not completed — Poor/non compliance on/after Week | 2 | 2
Not completed — No longer meets criteria on/after Wk 48 | 2 | 2
Not completed — Pregnancy on/after Week 48 | 1 | 2
Not completed — Withdrew consent on/after Week 48 | 0 | 2
Not completed — Continuing treatment | 385 | 368
Not completed — Lost to follow-up on/after Week 48 | 0 | 3
Not completed — Never treated | 2 | 3
Period: Baseline Through Week 96
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Started | 440 (Number randomized to ATV) | 443 (Number randomized to LPV)
RECEIVED ANY TREATMENT | 441 (1 participant randomized to LPV received ATV instead (treatment error)) | 437 (3 participants received ATV instead of LPV (treatment error) and 3 participants never treated)
Completed | 301 | 307
Not Completed | 139 | 136
Not completed — Adverse event before Week 96 | 13 | 22
Not completed — Death before Week 96 | 6 | 5
Not completed — Lack of efficacy before Week 96 | 16 | 10
Not completed — Lost to follow up before Week 96 | 10 | 13
Not completed — Participant Imprisoned before Week 96 | 1 | 0
Not completed — Poor/non compliance before Week 96 | 12 | 16
Not completed — Pregnancy before Week 96 | 5 | 7
Not completed — No longer meets criteria before Week 96 | 4 | 3
Not completed — Withdrew consent before Week 96 | 5 | 18
Not completed — Changed address before Week 96 | 0 | 1
Not completed — Lost to follow-up at Week 96 | 1 | 0
Not completed — Poor/non compliance at Week 96] | 2 | 0
Not completed — Pregnancy at Week 96 | 1 | 0
Not completed — Never treated | 2 | 3
Not completed — Continuing on treatment | 61 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD | Total
Number analyzed (Participants) | 440 | 443 | 883
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (9.1) | 37 (10.0) | 36 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 139 | 277
  Male | 302 | 304 | 606
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 42 | 41 | 83
  Black or African American | 83 | 80 | 163
  White | 207 | 221 | 428
  Hispanic/Latino | 7 | 6 | 13
  Mestizo | 71 | 68 | 139
  Mixed race | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human-immunodeficiency Virus- Ribonucleic Acid (HIV-RNA) < 50 Copies (c)/mL at Week 48
Description: HIV RNA < 50 c/mL is the most stringent measure of viral suppression (lowest threshold of assay) and indicates that a participant responded to treatment.
Time Frame: Baseline (Day 1) and Week 48
Population: Intent-to-treat (ITT) analysis. Participants received treatment assignment from the central randomization center. In this analysis, participants who did not complete the study were counted as having failed to respond to treatment. Participants who discontinued prior to obtaining Week 48 HIV RNA levels were categorized under non-completers.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 440 | 443
Participants | 343 | 338
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Treatment regimens compared by calculation of the difference in proportions (atazanavir/ritonavir- lopinavir/ritonavir) and 95% CI based on stratified normal approximation.Analyses were stratified by the same strata as randomization-HIV RNA level at enrollment and geographic region.The proportion of participants with HIV RNA below 50 copies/mL was computed within each stratum, and combined by use of a weighted average with weights proportional to stratum size:Cochran-Mantel-Haenszel weighting; Test type: Superiority or Other; Cochran-Mantel-Haenszel — Assuming 70% response rate (70% of participants remain on treatment for 48 wks and HIV RNA <50 copies/mL) on both regimens, sample size of 882 randomized participants (441/regimen) provided 90% power to demonstrate ATV/RTV is non-inferior to LPV/RTV; The ATV/RTV regimen was deemed to be non-inferior to the lopinavir/ritonavir regimen if the lower CI for the difference in proportions > -10%; Difference Estimate = 1.7, 95% CI 2-sided [-3.8 to 7.1]

2. Secondary Outcome: Number of Participants With HIV RNA < 400 c/mL at Week 48
Description: HIV RNA < 400 c/mL is a less stringent measure of viral suppression (highest threshold of assay) and indicates that a participant responded to treatment.
Time Frame: Baseline (Day 1) and Week 48
Population: Efficacy analyses of the treatment period are based on randomized population. In this analysis, participants who did not complete the study are counted as having failed to respond to treatment. Participants who discontinued prior to obtaining Week 48 HIV RNA levels were categorized under Non-completers.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 440 | 443
Participants | 377 | 365
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Treatment regimens were compared by calculation of the difference in proportions (ATV/RTV-LPV/RTV) and 95% CI based on a stratified normal approximation. Analyses were stratified by the same strata as randomization-ie, HIV RNA level at enrollment and geographic region. The proportion of participants with HIV RNA below 400 copies per mL was computed within each stratum, and combined by use of a weighted average with weights proportional to stratum size (Cochran-Mantel-Haenszel weighting); Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference Estimate = 3.3, 95% CI 2-sided [-1.5 to 8.1]

3. Secondary Outcome: Number of Participants With Confirmed Plasma HIV RNA < 400 c/mL at Week 48 (Defined by the Food and Drug Administration [FDA] Time to Loss of Virologic Response [TLOVR] Algorithm)
Description: TLOVR defines responders at Week 48 as participants with confirmed HIV RNA <400 c/mL through Week 48 without intervening virologic rebound or treatment discontinuation. Virologic rebound is defined as confirmed on-treatment HIV RNA <400 c/mL or last on-treatment HIV RNA <400 c/mL followed by discontinuation. Participants are considered failures in this analysis if they experienced virologic rebound at or before Week 48, discontinued before Week 48, never responded by Week 48, never received study therapy or had missing HIV RNA at Week 48 and beyond.
Time Frame: Baseline (Day 1) and Week 48
Population: Efficacy analyses of the treatment period are based on randomized population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 440 | 443
Participants | 377 | 363

4. Secondary Outcome: Reduction of log10 HIV RNA Levels From Baseline to Week 48
Description: Changes from baseline in log10 HIV RNA levels were calculated.
Time Frame: Baseline (Day 1) and Week 48
Population: All treated participants with data for this parameter.
Measure: Mean (Standard Error); unit: c/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 397 | 379
c/mL | -3.09 (0.042) | -3.13 (0.037)

5. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Count at Week 48
Description: Mean change from baseline in CD4 cell counts was determined.
Time Frame: Baseline (Day 1) and Week 48.
Population: All treated participants with data for this parameter.
Measure: Mean (Standard Error); unit: c/mm^3
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 370 | 363
c/mm^3 | 203 (7.1) | 219 (7.2)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Mean changes in CD4 cell counts from baseline at week 48 were compared between treatment regimens with 95% CIs based on stratified normal approximations and observed values; Test type: Superiority or Other; 95% CI comparison of difference; Difference Estimate = -16.4, 95% CI 2-sided [-35.9 to 3.1]

6. Secondary Outcome: Treatment Emergent Resistance in Isolates From Participants With Virologic Failure at Week 48
Description: Participants with virologic failure are those who never suppressed (HIV RNA <400 c/mL) and were on study through Week 48, or who rebounded to HIV RNA >= 400 c/mL and those who discontinued due to insufficient viral load response. IAS=International AIDS Society, PI=protease inhibitor, RTI=reverse transcription inhibitor, TAMS=Thymidine Analogue-Associated Mutations, NRTI=non-nucleotide reverse transcriptase inhibitor, M184V= Methionine-to-valine mutation at position 184 (in reverse transcription [RT] gene), FC=fold change
Time Frame: Baseline (Day 1) and Week 48
Population: Paired baseline and on-study HIV samples tested for genotypic resistance and phenotypic resistance. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 440 | 443
Participants
  Virologic Failure, Week 48 (HIV RNA >= 400 c/mL) | 27 | 26
  Paired Genotypes (n = 27, 26) | 17 | 15
  Paired Phenotypes (n= 27, 26) | 18 | 16
  IAS-defined major PI substitutions (n = 17, 15) | 1 | 0
  Other IAS-defined PI substitutions (n = 17, 15) | 6 | 2
  PI phenotypic resistance (ATV/RTV FC>5.2 (n=18,16) | 1 | 0
  PI phenotypic resistance (LPV/RTV FC >9 (n=18, 16) | 0 | 0
  PI phenotypic resistance (Other PIs )(n=18, 16) | 4 | 4
  RTI Substitutions , TAMS (n= 17,15) | 1 | 1
  RTI Substitutions , M184V (n = 17,15) | 3 | 3
  RTI phenotypic resistance, FTC FC>3.5 (n = 18, 16) | 4 | 3
  RTI phenotypic resistance, TDF FC >1.4(n = 18, 16) | 0 | 1
  RTI phenotypic resistance, Other NRTIs(n = 18, 16) | 5 | 5

7. Secondary Outcome: Number of Participants Who Died, Experienced Other Serious Adverse Events (SAEs), Experienced Adverse Events (AEs) and Experienced AEs Leading to Discontinuation Through Week 48
Description: AEs:new,untoward medical occurrences/worsening of pre-existing medical condition,drug-related or not.SAEs:any AE that:resulted in death;was life threatening;resulted in a persistent or significant disability/incapacity;resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; was cancer;or overdose.Discontinuation from study was due either to an AE or was conducted at the investigator's discretion.AEs represented here include SAEs, which are not included in the AE count represented in the AE xml upload section. As such, these numbers may not match.
Time Frame: From baseline (Day 1) to Week 48.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Deaths | 6 | 6
  Other SAEs | 51 | 42
  AEs | 400 | 399
  AEs leading to discontinuation | 11 | 15

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Hematology Through Week 48: Hemoglobin, Hematocrit, Platelet Count, International Normalized Ratio (INR), Neutrophils, Prothrombin Time (PT) and White Blood Cells (WBC)
Description: Hematology abnormalities were graded per modified World Health Organization (WHO) criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe). Grade 3 and 4 criteria were: Hemoglobin: Grade 3: 6.5-7.9 g/dL, Grade 4: <6.5 g/dL; Hematocrit: Grade 3: >=19.5 - 24%, Grade 4: <19.5%; platelet count: Grade 3: 20,000- 49, 999/ mm^3, Grade 4: <20,000/mm^3; INR: Grade 3 Absolute Neutrophil Count (ANC): Grade 3: >= 500 - <750/mm^3, Grade 4: <500/mm^3; PT: Grade 3: 1.51 - 3.0*ULN, Grade 4: >3*ULN; WBC: Grade 3: >=800 to <1000/mm^3, Grade 4: <80/mm^3.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: Safety analyses of the treatment period are based on treated population. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Hematocrit (n= 434, 431) | 0 | 6
  Hemoglobin (n= 434, 431) | 2 | 6
  INR (n= 435, 431) | 6 | 11
  Neutrophils (n = 434, 431) | 14 | 3
  Platelets ( n= 433, 430) | 5 | 1
  PT (n = 435, 431) | 6 | 16
  WBC (n = 434, 431) | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Serum Enzymes Levels Through Week 48
Description: Laboratory measurements marked as abnormal, as per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe). Grade 3 and 4 criteria in serum enzymes were: Creatine phosphokinase (CPK): Grade 3: 5.1 - 10.0 * upper limit of normal (ULN), Grade 4: >10* ULN; Lipase: Grade 3: 2.10 - 5.0* ULN, Grade 4: 5.0* ULN.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: Safety analyses of the treatment period are based on treated population.The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  CPK (n = 435, 430) | 22 | 20
  Lipase (n = 435, 430) | 6 | 6

10. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Liver Function Test Through Week 48
Description: Liver function tests abnormalities were graded as per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe), while albumin was graded as per National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE). Grade 3 and 4 criteria were: alanine aminotransferase (ALT), aspartate aminotransferase(AST), alkaline phosphatase: Grade 3: 5.1- 10*ULN, Grade 4: >10*ULN; direct and total bilirubin: Grade 3: 2.6- 5*ULN, Grade 4: >5*ULN, Albumin: Grade 3: <2g/dL.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  ALT (n= 435, 431) | 8 | 6
  AST (n = 435, 430) | 9 | 2
  Albumin (n = 435, 431) | 0 | 0
  Alkaline Phosphatase (n= 435, 430) | 1 | 1
  Direct Bilirubin (n = 435, 430) | 37 | 4
  Total Bilirubin (n = 435, 431) | 146 | 1

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Renal Function Test Through Week 48
Description: Renal function test abnormalities were graded as per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe). Grade 3 and 4 criteria were: Blood urea nitrogen (BUN): Grade 3: 5.1- 10*ULN, Grade 4: >10*ULN; Creatinine: Grade 3: 3.1 - 6*ULN, Grade 4: >6*ULN; low phosphorous (hypophosphatemia): Grade 3: 1.0- 1.4 mg/dL, Grade 4: <1.0mg/dL; high uric acid (hyperuricemia): Grade 3: 12.1 - 15.0 mg/dL, Grade 4: >15.0 mg/dL.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  BUN (n = 435, 431) | 0 | 0
  Creatinine (n = 435, 431) | 1 | 1
  Phosphorus (n = 435, 431) | 0 | 1
  Uric acid (n = 435, 431) | 0 | 3

12. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Electrolytes Through Week 48
Description: Serum electrolytes abnormalities,graded per modified WHOcriteria.Ranges were:hypercarbia:Grade3:41-45milliequivalents(meq)/L,Grade4:>45meq/L;hypocarbia:Grade3:10-14 meq/L,Grade4:<10 meq/L;hypercalcemia:Grade3:12.6 - 13.5 mg/dL,Grade 4:>13.5 mg/dL;hypocalcemia:6.1-6.9mg/dL,Grade4:<6.1mg/dL;hyperchloremia:Grade 3: 121-125 meq/L,Grade4:>125meq/L;hypochloremia:Grade 3:80-84 meq/L,Grade4:<80meq/L;hyperkalemia:Grade3:6.6-7.0meq/L,Grade4:>7.0meq/L;hypokalemia:Grade3:2.0-2.4 meq/L,Grade4:<2.0meq/L;hypernatremia:Grade3:158-165 meq/L,Grade4:>165meq/L;hyponatremia:Grade 3:116-122 meq/L,Grade 4:115 meq/L.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Hypercarbia (n = 435, 431) | 0 | 0
  Hypocarbia (n = 435, 431) | 1 | 7
  Hypercalcemia (n = 435, 431) | 0 | 0
  Hypocalcemia (n = 435, 431) | 1 | 4
  Hyperchloremia (n = 435, 431) | 0 | 0
  Hypochloremia (n = 435, 431) | 0 | 0
  Hyperkalemia (n = 435, 430) | 0 | 1
  Hypokalemia (n = 435, 430) | 0 | 1
  Hypernatremia (n = 435, 431) | 0 | 0
  Hyponatremia (n = 435, 431) | 0 | 1

13. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Urinalysis Through Week 48
Description: Laboratory measurements marked as abnormal, per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe), at any study time point. The following Grade 3 and 4 definitions specify the criteria for MAs in urinalysis: Proteinuria: Grade 3: 4= or >2-3.5 g loss/day, Grade 4: >3.5 g loss/day.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Glycosuria (n = 434, 431) | 4 | 3
  Proteinuria (n = 434, 431) | 3 | 1

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Fasting Lipids Through Week 48
Description: Laboratory measurements marked as abnormal, as per National Cholesterol Education Program (NCEP)- Adult Treatment Panel (ATP)-III guided categories. The following definitions specify the criteria for MAs in fasting lipids: Total cholesterol: Grade 3: 240 - 300 mg/dL, Grade 4: >=240 mg/dL, triglycerides: Grade 3: 200 - <500 mg/dL, Grade 4: >=500 mg/dL.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Total Cholesterol (n = 434, 428) | 30 | 77
  Triglycerides (n = 434, 428) | 2 | 15

15. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Fasting Glucose Through Week 48
Description: Laboratory measurements marked as abnormal, per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe), at any study time point. The following Grade 3 and 4 definitions specify the criteria for MAs in fasting glucose: hypoglycemia: Grade 3: 30-39 mg/dL, Grade 4: <30 mg/dL; hyperglycemia: 251-500 mg/dL, Grade 4: >500 mg/dL.
Time Frame: At Screening (Day -30), Baseline (Day 1), Week 4, 12, 24, 36, and 48.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Hyperglycemia (n = 434, 428) | 1 | 1
  Hypoglycemia (n = 434, 428) | 0 | 0

16. Secondary Outcome: Mean Change in Weight From Baseline at Week 48
Description: Mean change in body weight from baseline was determined.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety analyses of the treatment period are based on treated population, who had values for this parameter.
Measure: Mean (Standard Error); unit: kg
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 395 | 370
kg | 4.0 (0.3) | 2.0 (0.3)

17. Secondary Outcome: Mean Change in Body Mass Index (BMI) in Participants at Week 48
Description: Mean change in BMI from baseline at Week 48 was determined.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety analyses of the treatment period are based on treated population, who had values for this parameter.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 393 | 370
kg/m^2 | 1.3 (0.10) | 0.8 (0.10)

18. Secondary Outcome: Mean Change in Fasting Lipid at Week 48
Description: Mean change from baseline in fasting lipids, for fasting total cholesterol, LDL cholesterol, HDL cholesterol, non-HDL cholesterol, and triglycerides at Week 48 were determined.
Time Frame: Baseline (Day 1) and Week 48.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
milligrams/deciliter (mg/dL)
  Fasting total Cholesterol (n=373, 337) | 19 (1.6) | 38 (1.8)
  Fasting HDL Cholesterol (n=371, 335) | 9 (0.6) | 12 (0.6)
  Fasting Non-HDL Cholesterol (n=371, 335) | 10 (1.5) | 26 (1.7)
  Fasting LDL Cholesterol (n=372, 335) | 12 (1.4) | 18 (1.5)
  Fasting Triglycerides (n=373, 337) | 20 (4.0) | 70 (5.7)

19. Secondary Outcome: Mean Change in Fasting Glucose at Week 48
Description: Mean change from baseline in fasting glucose at Week 48.
Time Frame: Baseline (Day 1) and Week 48.
Population: Safety analyses of the treatment period are based on treated population with values for this parameter.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 383 | 363
mg/dL | 2 (0.6) | 0 (1.3)

20. Secondary Outcome: Mean Change in Fasting Insulin at Week 48
Description: Mean change from baseline in fasting insulin at Week 48.
Time Frame: Baseline (Day 1) and Week 48.
Population: Safety analyses of the treatment period are based on treated population with values for this parameter.
Measure: Mean (Standard Error); unit: micro units (µU)/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 371 | 352
micro units (µU)/mL | 2.5 (0.52) | 0.2 (0.38)

21. Secondary Outcome: Mean Change From Baseline in Quality of Life as Measured by the Medical Outcomes Survey - Human Immunodeficiency Virus (MOS-HIV) at Week 24
Description: Medical Outcomes Study HIV Health Survey (MOS-HIV) is developed to assess a patient's health and functional status associated with HIV infection. The MOS-HIV questionnaire is applied to participants with adequate linguistic skills. The subscale and summary scores range from 0-100 with a higher score indicating better health.
Time Frame: Baseline (Day 1) and Week 24.
Population: As-treated participants with evaluable baseline MOS-HIV . The 'n' is signifying those participants who were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 347 | 351
Units on Scale
  Physical Health Summary (317, 314) | 4.1 (0.46) | 3.3 (0.46)
  Mental Health Summary (317, 314) | 5.3 (0.50) | 4.8 (0.52)
  Overall Health Perception Subscale (325, 320) | 15.2 (1.31) | 13.0 (1.41)
  Physical Function Subscale (324, 325) | 7.6 (1.25) | 5.0 (1.30)
  Role Function Subscale (325, 325) | 10.6 (1.72) | 6.5 (1.61)
  Social Function Subscale (327, 322) | 8.5 (1.54) | 7.1 (1.49)
  Cognitive Function Subscale (326, 324) | 5.6 (1.11) | 3.0 (0.94)
  Pain Subscale (327, 325) | 7.4 (1.37) | 8.6 (1.23)
  Mental Health Subscale (325, 326) | 6.4 (1.09) | 7.4 (1.08)
  Energy/Fatigue Subscale (323, 326) | 7.1 (1.16) | 7.5 (1.14)
  Health Distress Subscale (323, 326) | 14.4 (1.29) | 13.9 (1.30)
  Quality of Life Subscale (327, 326) | 9.9 (1.32) | 7.1 (1.29)
  Health Transition Subscale (327, 326) | 13.1 (1.64) | 10.7 (1.55)

22. Secondary Outcome: Mean Change From Baseline in Quality of Life as Measured by the Medical Outcomes Survey - Human Immunodeficiency Virus (MOS-HIV) at Week 48
Description: MOS-HIV is developed to assess a participant's health and functional status associated with HIV infection. The questionnaire is applied to participants with adequate linguistic skills and consists of 35 items. The questionnaire derives an overall health score and 10 subscale scores (health transitions, pain, physical functioning, role functioning, social functioning, cognitive functioning, mental health, energy/fatigue, health distress and quality of life).The subscale and summary scores range from 0-100 with a higher score indicating better health.
Time Frame: Baseline (Day 1) and Week 48
Population: Participants analyzed are as-treated participants with evaluable baseline MOS-HIV. The 'n' is signifying those participants who were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 347 | 351
Units on Scale
  Physical Health Summary (296, 287) | 3.8 (0.50) | 3.3 (0.49)
  Mental Health Summary (296, 287) | 6.0 (0.54) | 5.6 (0.54)
  Overall Health Perception Subscale (305, 297) | 15.6 (1.53) | 13.7 (1.51)
  Physical Function Subscale (303, 298) | 5.8 (1.28) | 5.3 (1.24)
  Role Function Subscale (307, 298) | 8.5 (1.75) | 8.1 (1.75)
  Social Function Subscale (308, 295) | 9.2 (1.48) | 7.4 (1.66)
  Cognitive Function Subscale (307, 300) | 4.8 (1.25) | 5.6 (1.05)
  Pain Subscale (308, 297) | 8.3 (1.39) | 8.0 (1.39)
  Mental Health Subscale (306, 300) | 8.3 (1.21) | 8.7 (1.10)
  Energy/Fatigue Subscale (304, 300) | 8.4 (1.25) | 7.9 (1.21)
  Health Distress Subscale (304, 300) | 14.3 (1.39) | 15.0 (1.36)
  Quality of Life Subscale (308, 300) | 12.9 (1.39) | 8.4 (1.34)
  Health Transition Subscale (308, 300) | 11.0 (1.63) | 8.8 (1.64)

23. Secondary Outcome: Mean Change From Baseline (BL) in Quality of Life as Measured by the Impact of Gastro-intestinal Toxicity at Week 4 (IBS-QoL)
Description: The IBS-QoL questionnaire has 34 items and an overall score and 8 subscale scores: dysphoria,interference with activity,body image,health worry, food avoidance,social reaction,sexual, and relationships. Overall and subscores transformed to a 0-100 scale (0=lowest score, 100=highest possible score). Scores between these values represent the percentage of the total possible score achieved. Higher scores=better IBS-related QoL. A 14-point change from BL in IBS-QoL score in women with moderate to severe functional bowel disorders is a minimally important difference based on pain and satisfaction.
Time Frame: IBS-QoL is administered at baseline (Day 1) and Week 4.
Population: As treated participants with evaluable baseline IBS-QOL. The 'n' is signifying those participants were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 343 | 349
Units on Scale
  Overall (306, 316) | 3.2 (0.71) | -0.7 (0.66)
  Dysphoria (317, 325) | 3.3 (0.79) | -0.1 (0.75)
  Interference with activity (319, 327) | 3.1 (0.86) | -1.9 (0.79)
  Body image (321, 329) | 1.6 (0.71) | -1.3 (0.68)
  Health worry (319, 330) | 6.0 (0.96) | 2.0 (0.99)
  Food avoidance (319, 329) | 4.0 (1.03) | -1.7 (1.07)
  Social reaction (316, 327) | 1.9 (0.76) | -0.8 (0.71)
  Sexual (320, 329) | 3.7 (1.06) | -0.1 (1.02)
  Relationships (321, 328) | 1.2 (0.72) | -0.6 (0.75)

24. Secondary Outcome: Mean Change From Baseline in Quality of Life as Measured by the Impact of Gastro-intestinal Toxicity at Week 12 (IBS-QoL)
Description: as for outcome 23
Time Frame: IBS-QoL is administered at baseline (Day 1) and Week 12.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 343 | 349
Units on Scale
  Overall (301. 310) | 4.6 (0.69) | 0.2 (0.89)
  Dysphoria (308, 319) | 4.7 (0.79) | 1.2 (0.94)
  Interference with activity (310, 320) | 5.1 (0.83) | -0.4 (0.96)
  Body image (316, 321) | 2.1 (0.69) | -0.1 (0.85)
  Health worry (312, 320) | 7.9 (1.02) | 3.6 (1.23)
  Food avoidance (316, 322) | 5.6 (0.95) | -0.6 (1.25)
  Social reaction (311, 316) | 3.3 (0.73) | -0.4 (0.95)
  Sexual (317, 321) | 4.7 (1.11) | -0.4 (1.19)
  Relationships (313, 320) | 3.5 (0.75) | 0.0 (0.99)

25. Secondary Outcome: Mean Change From Baseline in Quality of Life as Measured by the Impact of Gastro-intestinal Toxicity at Week 24 Using the Irritable Bowel Syndrome Quality of Life (IBS-QoL)
Description: as for outcome 23
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 343 | 349
Units on a scale
  Overall (290, 289) | 4.3 (0.77) | 1.4 (0.88)
  Dysphoria (295, 298) | 4.4 (0.84) | 1.8 (0.97)
  Interference with activity (294, 297) | 4.4 (0.92) | 0.0 (1.04)
  Body image (299, 300) | 1.8 (0.80) | 1.1 (0.84)
  Health worry (297, 300) | 7.5 (0.99) | 5.3 (1.18)
  Food avoidance (299, 300) | 5.6 (1.14) | 0.4 (1.29)
  Social reaction (295, 297) | 3.2 (0.80) | 0.4 (0.92)
  Sexual (299, 299) | 4.3 (1.20) | 0.8 (1.15)
  Relationships (297, 297) | 3.3 (0.89) | 1.2 (1.00)

26. Secondary Outcome: Number of Participants Who Adhered to Regimen as Measured by Multicenter AIDS Cohort Study Adherence Questionnaire (MACS) at Week 48
Description: The MACS adherence questionnaire asks patients how many medication doses they missed during the previous day, 2 days, 3 days and 4 days. Adherence to regimen was defined as taking 100% of medicine (all doses and numbers of pills as prescribed for each medicine). This strict adherence cut-off was based on the guidelines stating that anything less than excellent adherence may result in a virus breakthrough and development of resistance.
Time Frame: Week 48
Population: The 'n' is signifying those participants who were evaluated for this measure at the timepoint for each group respectively.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 401 | 378
Participants | 330 | 316

27. Secondary Outcome: Number of Participants With HIV RNA < 50 c/mL) at Week 96
Description: HIV RNA < 50 c/mL is the most stringent measure of viral suppression (lowest threshold of assay) and indicates that a participant has responded to treatment.
Time Frame: Baseline (Day 1) and Week 96
Population: Efficacy analyses of the treatment period are based on randomized population. In this analysis, participants who did not complete the study are counted as having failed to respond to treatment. Participants who discontinued prior to obtaining Week 96 HIV RNA levels were categorized under Non-completers.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 440 | 443
Participants | 327 | 302
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cochran-Mantel-Haenszel — Assuming 70% response rate (70% of participants remain on treatment for 96 wks and HIV RNA <50 copies/mL) on both regimens, sample size of 882 randomized participants (441/regimen) provided 90% power to demonstrate ATV/RTV is non-inferior to LPV/RTV; [statistical method as in outcome 1, analysis 1]; Difference Estimate = 6.1, 95% CI 2-sided [0.3 to 12.0]

28. Secondary Outcome: Number of Participants With HIV RNA < 400 c/mL) at Week 96
Description: HIV RNA <400 c/mL is a less stringent measure of viral suppression (highest threshold of assay) and indicates that a participant has responded to treatment.
Time Frame: Baseline (Day 1) and Week 96
Population: as for outcome 27
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 440 | 443
Participants | 350 | 330
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Difference Estimate = 5.1, 95% CI 2-sided [-0.4 to 10.6]

29. Secondary Outcome: Reduction of log10 HIV RNA Levels From Baseline at Week 96
Description: Changes from baseline in log10 HIV RNA levels were calculated.
Time Frame: Baseline (Day 1) and Week 96
Population: Efficacy analyses of the treatment period are based on as-randomized population with values for this parameter. log10 HIV RNA changes from baseline were summarized at Week 96 using observed values.
Measure: Mean (Standard Error); unit: c/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 360 | 340
c/mL | -3.21 (0.034) | -3.19 (0.036)

30. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at Week 96
Description: Mean change from baseline in CD4 count among treated participants was determined.
Time Frame: Baseline (Day 1) and Week 96
Population: Efficacy analyses of the treatment period are based on as-randomized population with values for this parameter.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 336 | 317
cells/mm^3 | 268 (7.6) | 290 (8.7)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; 95% CI comparison of difference; Difference Estimate = -21.2, 95% CI 2-sided [-43.3 to 0.9]

31. Secondary Outcome: Number of Participants Who Died, Experienced Other Serious Adverse Events (SAEs), Experienced Adverse Events (AEs) and Experienced Events Leading to Discontinuation Through Week 96
Description: as for outcome 7
Time Frame: From Day 1 through Week 96
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Deaths | 6 | 6
  Serious Adverse Events (SAEs) | 63 | 50
  Adverse Events (AEs) leading to discontinuation | 13 | 22

32. Secondary Outcome: Mean Changes in Fasting Lipids at Week 96
Description: Mean change from baseline in fasting lipids at Week 96 was determined.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
mg/dL
  Fasting total Cholesterol (n=342, 291) | 20 (1.8) | 37 (1.8)
  Fasting HDL Cholesterol (n=341, 291) | 7.0 (0.6) | 10.0 (0.7)
  Fasting Non-HDL Cholesterol (n=341, 291) | 13.0 (1.6) | 27.0 (1.7)
  Fasting LDL Cholesterol (n=342, 291) | 12.0 (1.5) | 17.0 (1.5)
  Fasting Triglycerides (n=342, 291) | 16.0 (4.4) | 63.0 (5.4)

33. Primary Outcome: Maximum Plasma Concentration (Cmax) of ATV/RTV and LPV/RTV in the Presence of an Antiretroviral (ARV) Regimen Including TDF at Week 4
Description: Cmax was derived from plasma concentration versus time data.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 Hrs post dosing with ATV/RTV and TDF all given every day (QD) and at predose, 1, 2, 3, 4, 6, 8, 12 Hrs post dosing with LPV/RTV given twice daily (BID) and TDF given QD.
Population: All participants who completed the intensive pharmacokinetic (PK) study.
Measure: Geometric Mean (Full Range); unit: nanogram(ng)/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
nanogram(ng)/mL | 2897 [837.0 to 5610] | 10654 [5658 to 31316]

34. Secondary Outcome: Mean Changes in Fasting Glucose at Week 96
Description: Mean change from baseline in fasting glucose at Week 96 was determined.
Time Frame: Baseline (Day 1) and Week 96
Population: Safety analyses of the treatment period are based on treated population with values for this parameter.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 355 | 330
mg/dL | 4.0 (1.2) | 1.0 (1.4)

35. Secondary Outcome: Mean Changes in Fasting Insulin at Week 96
Description: Mean change from baseline in fasting insulin at Week 96.
Time Frame: Baseline (Day 1) and Week 96.
Population: Safety analyses of the treatment period are based on treated population with values for this parameter.
Measure: Mean (Standard Error); unit: µU/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 349 | 324
µU/mL | 0.1 (0.47) | -0.8 (0.43)

36. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Hematology: Hemoglobin, Hematocrit, Platelet Count, INR, Neutrophils, PT and WBC Through Week 96
Description: Hematology abnormalities were graded per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe). Grade 3 and 4 criteria were: Hemoglobin: Grade 3: 6.5-7.9 g/dL, Grade 4: <6.5 g/dL; Hematocrit: Grade 3: >=19.5 - 24%, Grade 4: <19.5%; platelet count: Grade 3: 20,000- 49, 999/ mm^3, Grade 4: <20,000/mm^3; INR: Grade 3 Absolute Neutrophil Count (ANC): Grade 3: >= 500 - <750/mm^3, Grade 4: <500/mm^3; PT: Grade 3: 1.51 - 3.0*ULN, Grade 4: >3*ULN; WBC: Grade 3: >=800 to <1000/mm^3, Grade 4: <80/mm^3.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Hematocrit (n= 434, 431) | 0 | 6
  Hemoglobin (n= 434, 431) | 3 | 7
  INR (n= 435, 431) | 7 | 18
  Neutrophils (n = 434, 431) | 21 | 7
  Platelets ( n= 433, 431) | 5 | 1
  Prothrombin time (n = 435, 431) | 9 | 24
  WBC (n = 434, 431) | 0 | 1

37. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Serum Enzyme Levels Through Week 96
Description: Laboratory measurements marked as abnormal, as per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe). Grade 3 and 4 criteria in serum enzymes were: CPK: Grade 3: 5.1 - 10.0 * ULN, Grade 4: >10* ULN; Lipase: Grade 3: 2.10 - 5.0* ULN, Grade 4: 5.0* ULN.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  CPK (n=435, 430) | 34 | 28
  Lipase (n=435, 430) | 9 | 9

38. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Liver Function Test Through Week 96
Description: Liver function tests abnormalities were graded as per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe), while albumin was graded as per NCI-CTCAE. Grade 3 and 4 criteria were: ALT, AST, alkaline phosphatase: Grade 3: 5.1- 10*ULN, Grade 4: >10*ULN; direct and total bilirubin: Grade 3: 2.6- 5*ULN, Grade 4: >5*ULN, Albumin: Grade 3: <2g/dL.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  ALT (n= 435, 431) | 11 | 7
  AST (n = 435, 430) | 11 | 5
  Albumin (n = 435, 431) | 0 | 0
  Alkaline Phosphatase (n= 435, 430) | 1 | 1
  Total Bilirubin (n = 435, 431) | 192 | 3

39. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Renal Function Test Through Week 96
Description: Renal function test abnormalities were graded as per modified WHO criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = very severe). Grade 3 and 4 criteria were: BUN: Grade 3: 5.1- 10*ULN, Grade 4: >10*ULN; Creatinine: Grade 3: 3.1 - 6*ULN, Grade 4: >6*ULN; low phosphorous (hypophosphatemia): Grade 3: 1.0- 1.4 mg/dL, Grade 4: <1.0mg/dL; high uric acid (hyperuricemia): Grade 3: 12.1 - 15.0 mg/dL, Grade 4: >15.0 mg/dL.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  BUN (n = 435,431) | 0 | 0
  Creatine (n = 435, 431) | 1 | 2
  Phosphorous (n = 435, 431) | 0 | 1
  Uric acid (n = 435, 431) | 1 | 4

40. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Electrolytes Level Through Week 96
Description: as for outcome 12
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Hypercarbia (n = 435, 431) | 0 | 0
  Hypocarbia (n = 435, 431) | 4 | 8
  Hypercalcemia (n = 435, 431) | 0 | 0
  Hypocalcemia (n = 435, 431) | 1 | 4
  Hyperchloremia (n = 435, 431) | 0 | 0
  Hypochloremia (n = 435, 431) | 0 | 2
  Hyperkalemia (n = 435, 430) | 0 | 1
  Hypokalemia (n = 435, 430) | 0 | 1
  Hypernatremia (n = 435, 431) | 1 | 2
  Hyponatremia (n = 435, 431) | 0 | 2

41. Primary Outcome: Area Under the Concentration-time Curve, in One Dosing Interval [AUC(TAU)] of ATV/RTV and LPV/RTV in the Presence of an ARV Regimen Including TDF at Week 4
Description: AUC(TAU) was derived from the plasma concentration versus time data. It was calculated from time 0 to 12 hours for LPV and RTV in the LPV/RTV regimen, 0-24 hours for ATV and RTV in the ATV/RTV regimen, and 0-24 hours for tenofovir in both regimens at Week 4.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 Hrs post dosing with ATV/RTV and TDF all given QD and at predose, 1, 2, 3, 4, 6, 8, 12 Hrs post dosing with LPV/RTV given BID and TDF given QD.
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
ng*h/mL | 28605 [9908 to 58872] | 90945 [43260 to 302989]

42. Primary Outcome: Minimum Plasma Concentration (Cmin) of ATV/RTV and LPV/RTV in the Presence of an ARV Regimen Including TDF at Week 4
Description: Cmin was derived from the plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
ng/mL | 526.4 [130.0 to 1350] | 5944 [1555 to 22739]

43. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of ATV/RTV and LPV/RTV in the Presence of an ARV Regimen Including TDF at Week 4
Description: Tmax was derived from the plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Median (Full Range); unit: Hr
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
Hr | 3.00 [1.50 to 24.00] | 4.00 [0.00 to 12.00]

44. Primary Outcome: Terminal Elimination Half-life (T-half) of ATV/RTV and LPV/RTV in the Presence of an ARV Regimen Including TDF at Week 4
Description: T-half was derived from the plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Mean (Standard Deviation); unit: Hr
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 17 | 12
Hr | 10.31 (3.32) | 13.89 (14.48)

45. Primary Outcome: Protein Binding Adjusted Effective Concentration (EC-90) of ATV and LPV When Dosed With RTV at Week 4
Description: EC90/50=concentration of drug inducing 90%/50% of its maximal response. Protein binding adjusted EC90 for ATV and LPV were derived from phenotypically measured individual EC50 values at baseline using the following formula: Protein binding adjusted EC90 (ng/mL) = scale factor × molecular weight of the free base × EC50 micrometer(μM)/ unbound fraction (fu). Scale factor relates EC50 to EC90 (value of 3 and 2 for ATV and LPV, respectively); fu: estimated unbound fraction of ATV and LPV in vivo (0.14 and 0.02 for ATV and LPV respectively).
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 17 | 19
ng/mL | 19.01 [8.29 to 35.23] | 162.7 [100.6 to 471.6]

46. Primary Outcome: Inhibitory Quotient (IQ) of ATV and LPV When Dosed With RTV at Week 4
Description: IQ defined as Cmin at week 4 divided by protein binding adjusted EC90 values for the respective protease inhibitor (ATV or LPV) derived from individual participant clinical isolates.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 17 | 19
ng/mL | 27.33 [3.94 to 77.27] | 35.91 [10.76 to 129.0]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 0.761, 90% CI 2-sided [0.507 to 1.142] — Point estimates and 90% confidence intervals (CIs) for differences between treatment regimens were calculated on the log scale, and were exponentiated to obtain estimates for ratios of geometric means on the original scale

47. Primary Outcome: Cmax of RTV at Week 4
Description: Cmax was derived from plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
ng/mL | 959.8 [139.0 to 2900] | 657.4 [193.8 to 1814]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 1.460, 90% CI 2-sided [1.005 to 2.121] — Point estimates and 90% CIs for differences between treatment regimens were calculated on the log scale, and were exponentiated to obtain estimates for ratios of geometric means on the original scale

48. Primary Outcome: AUC (0-24) of RTV at Week 4
Description: AUC (0-24) was derived from plasma concentration versus time data. It was estimated as 2 times the AUC(TAU) based on 12-hour PK.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
ng*h/mL | 6724 [1371 to 23854] | 8011 [2815 to 19929]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 0.839, 90% CI 2-sided [0.612 to 1.151] — [estimate comment as in outcome 47, analysis 1]

49. Primary Outcome: Cmin of RTV at Week 4
Description: Cmin was derived from plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 18 | 21
ng/mL | 50.52 [14.50 to 298.0] | 179.0 [42.82 to 763.8]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 0.282, 90% CI 2-sided [0.181 to 0.439] — [estimate comment as in outcome 47, analysis 1]

50. Primary Outcome: Cmax of Tenofovir at Week 4
Description: Cmax was derived from plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 17 | 20
ng/mL | 352.0 [104.8 to 641.8] | 380.7 [118.0 to 1801]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 0.925, 90% CI 2-sided [0.699 to 1.223] — [estimate comment as in outcome 47, analysis 1]

51. Primary Outcome: Cmin of Tenofovir at Week 4
Description: Cmin was derived from plasma concentration versus time data.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 17 | 20
ng/mL | 72.46 [21.08 to 114.7] | 84.98 [44.27 to 757.2]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 0.853, 90% CI 2-sided [0.626 to 1.161] — [estimate comment as in outcome 47, analysis 1]

52. Primary Outcome: AUC (TAU) of Tenofovir at Week 4
Description: AUC (TAU) was derived from plasma concentration versus time data.It was calculated from time 0-24 hours for tenofovir in LPV/RPV and ATV/RTV regimen at Week 4.
Time Frame: as for outcome 41
Population: All participants who completed the intensive PK study.
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 17 | 20
ng*h/mL | 3272 [1678 to 5486] | 3675 [2240 to 25385]
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Test type: Superiority or Other; ANOVA; point estimate = 0.890, 90% CI 2-sided [0.689 to 1.151] — [estimate comment as in outcome 47, analysis 1]

53. Primary Outcome: Mean Change From Baseline in Trunk-to-Limb Fat Ratio as Measured by Dual Energy X-ray Absorptiometry (DEXA) at Week 96
Description: Mean changes from baseline in trunk-to-limb fat ratio as measured by DEXA, an x-ray scan used to measure bone mineral density. Clinical improvement is associated with a decrease in values.
Time Frame: Baseline (Day 1) and Week 96.
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 106 | 70
Ratio | 0.05 (0.015) | 0.00 (0.015)

54. Primary Outcome: Number of Participants With Single Nucleotide Polymorphisms (SNPs) Included in Genotype-Phenotype Analysis
Description: 19 genes of interest were selected from previous results or literature, and 34 SNPs were genotyped. Phenotype-Genotype analysis was performed using 31 of the SNPs. The genotypes of each SNP were further classified as either a minor allele carrier (MAC) group composed of heterozygous and rare homozygous genotypes, or wild type [WT, common homozygous].
Time Frame: Baseline visit
Population: Participants with both genotypes and phenotypes available in the metabolic substudy. Phenotypes used in this analysis were from 3 time points: baseline (Week 0), Week 48, and Week 96. The Hardy-Weinberg Equilibrium test was used to check for the genotype quality. All SNPs passed the quality check.
Measure: Number; unit: participants
Groups:
- All Participants With Pharmacogenetic Blood Samples: Participants were administered an oral dose of Atazanavir (ATV) 300 mg and ritonavir (RTV) 100 mg once daily along with food. Doses were taken 24 hours apart at the same time as fixed dose combination tenofovir (TDF) 300 mg plus emtricitabine (FTC) 200 mg once daily.
Arm/Group | All Participants With Pharmacogenetic Blood Samples
Number analyzed (Participants) | 199
participants
  RETN_097 WT | 164
  RETN_097 MAC | 35
  APOE_R176C WT | 182
  APOE_R176C MAC | 16
  CCDC122_5980 WT | 126
  CCDC122_5980 MAC | 71
  IL6_5309 WT | 57
  IL6_5309 MAC | 141
  RS11030679 WT | 112
  RS11030679 MAC | 87
  APOE_C130R WT | 169
  APOE_C130R MAC | 30
  RETN_2265 WT | 146
  RETN_2265 MAC | 53
  RETN_598 WT | 119
  RETN_598 MAC | 80
  RETN_734 WT | 175
  RETN_734 MAC | 22
  BRUNOL_1842 WT | 121
  BRUNOL_1842 MAC | 77
  RETN_730 WT | 99
  RETN_730 MAC | 100

55. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Fasting Lipids Level Through Week 96
Description: Laboratory measurements marked as abnormal, as per NCEP-ATP-III guided categories. The following definitions specify the criteria for MAs in fasting lipids: Total cholesterol: Grade 3: 240 - 300 mg/dL, Grade 4: >=240 mg/dL, triglycerides: Grade 3: 200 - <500 mg/dL, Grade 4: >=500 mg/dL.
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Total Cholesterol (n = 434, 428) | 47 | 108
  Triglycerides (n = 434, 428) | 3 | 18

56. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Fasting Glucose Levels Through Week 96
Description: as for outcome 15
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Hyperglycemia (n = 434, 428) | 3 | 2
  Hypoglycemia (n = 434, 428) | 1 | 0

57. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Urinalysis Through Week 96
Description: as for outcome 13
Time Frame: At screening (Day -30), baseline (Day 1), Week 4, 12, 24, 36, 48, 60, 72, 84 and 96.
Population: Safety analyses of the treatment period are based on treated population.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 441 | 437
Participants
  Glycosuria (n = 434, 431) | 6 | 5
  Proteinuria (n = 434, 431) | 5 | 6

58. Secondary Outcome: Number of Participants With Virologic Failure Showing Treatment Emergent Resistance Through Week 96
Description: Virologic failure participants defined as participants who were never suppressed (HIV RNA < 400 c/mL) and on study through Week 48, or who rebounded to HIV RNA ≥ 400 c/mL, and those who discontinued due to insufficient viral load response using CVR (NC=F). IAS-USA=International AIDS Society-United States of America, PI=protease inhibitor, RTI=reverse transcription inhibitor, TAMS=Thymidine Analogue-Associated Mutations, NRTI=non-nucleotide reverse transcriptase inhibitor, M184/V= Methionine-to-valine mutation at position 184 (in reverse transcription [RT] gene), FC=fold change
Time Frame: Baseline (Day 1) and Week 96.
Population: Resistance analysis are based on randomized population. 2 subjects with baseline phenotypic resistance to ATV/RTV are excluded. Paired baseline and on-study HIV samples tested for genotypic resistance and phenotypic resistance. "n" signifies the number of participants evaluable for each parameter.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 438 | 443
Participants
  Virologic Failure, Week 96 (HIV RNA >= 400 c/mL) | 28 | 29
  Paired Genotypes (n = 28, 29) | 26 | 26
  Paired Phenotypes (n= 28, 29) | 25 | 23
  IAS-USA major PI substitutions (n = 26, 26) | 1 | 0
  IAS-USA minor PI substitutions (n = 26, 26) | 1 | 1
  PI polymorphisms without IAS-USA (n=26, 26) | 11 | 14
  PI phenotypic resistance (ATV/RTV FC >5.2 (25, 23) | 1 | 0
  PI phenotypic resistance (LPV/RTV FC>9 (25,23) | 0 | 1
  PI phenotypic resistance (Other PIs [25, 23]) | 3 | 6
  NRTI substitutions (TAMS [26, 26]) | 1 | 3
  NRTI substitutions (M184I/V [26, 26]) | 5 | 7
  RTI phenotypic resistance (FC [n = 25, 23]) | 5 | 5
  RTI phenotypic resistance (TDF [n = 25, 23]) | 0 | 2
  RTI phenotypic resistance (Other NRTI [n =25, 23]) | 5 | 6

59. Secondary Outcome: Mean Change From Baseline in Trunk-to-limb Fat Ratio Measured by DEXA at Week 48
Description: Mean changes from baseline in trunk-to-limb fat ratio as measured by DEXA, an x-ray scan used to measure bone mineral density. Clinical improvement was associated with a decrease in values.
Time Frame: DEXA scans were taken at Baseline (Day 1) and at Weeks 48.
Population: As-treated participants (with values for this parameter)in the lipodystrophy substudy who participated in the substudy and signed the informed consent for the substudy.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 118 | 81
Ratio | 0.04 (0.013) | -0.02 (0.014)

60. Secondary Outcome: Mean Percent Changes From Baseline in Limb, Trunk and Total Body Fat Measured by DEXA at Week 48
Description: The mean percent change from baseline in limb, trunk and total body fat was measured by DEXA. Limb fat: a physical sign of lipoatrophy, clinical improvement in limb fat is associated with a decrease in values. Trunk fat: a physical sign of lipohypertrophy, clinical improvement in trunk fat is associated with a decrease in values. Total body fat: association of many factors like trunk fat, limb fat, weight etc. Clinical improvement in total body fat cannot be predicted based solely an increase or decrease of these values.
Time Frame: DEXA scans were performed at baseline (within 30 days of starting study treatment), and at Weeks 48.
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 118 | 82
Percentage
  Trunk Fat | 26 [18.9 to 34.5] | 16 [9.4 to 22.2]
  Limb Fat | 22 [15.7 to 28.9] | 17 [11.2 to 23.1]
  Total Body Fat | 23 [16.7 to 29.9] | 15 [9.8 to 21.1]

61. Secondary Outcome: Mean Percent Changes From Baseline in Limb, Trunk and Total Body Fat Measured by DEXA at Week 96
Description: The mean percent change from baseline in limb, trunk and total body fat was measured by DEXA. Limb fat: a physical sign of lipoatrophy, clinical improvement in limb fat is associated with a decrease in values. Trunk fat: physical sign of lipohypertrophy, clinical improvement in trunk fat is associated with a decrease in values. Total body fat: association of many factors like trunk fat, limb fat, weight etc. Clinical improvement in total body fat cannot be predicted based solely an increase or decrease of these values.
Time Frame: Baseline (Day 1) and Week 96.
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 106 | 71
Percentage
  Trunk Fat | 34 [23.9 to 44.8] | 16 [8.0 to 24.0]
  Limb Fat | 27 [18.7 to 36.3] | 15 [8.3 to 22.6]
  Total Body Fat | 29 [20.5 to 38.3] | 15 [8.0 to 22.2]

62. Secondary Outcome: Median Changes From Baseline at Week 96 in VAT-to-TAT, VAT-to-SAT and, Trunk-to-limb Fat Ratio Measured by Computed Tomography (CT)/DEXA
Time Frame: Baseline (Day 1) and Week 96.
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy.
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 125 | 99
Ratio
  VAT-to-TAT Ratio (n = 95,68) | -0.04 [-0.06 to -0.02] | -0.02 [-0.04 to 0.00]
  VAT-to-SAT Ratio (n = 95, 68) | -0.22 [-0.41 to -0.04] | -0.09 [-0.18 to 0.00]
  Trunk-to-Limb Fat Ratio (n = 106, 71) | 0.05 [0.02 to 0.08] | 0.00 [-0.03 to 0.03]

63. Secondary Outcome: Mean Percent Changes From Baseline in Bone Mineral Density (BMD) Measured by DEXA at Week 48
Description: Mean percent change from baseline in BMD of arms, legs, trunk and total body was measured using DEXA, an X-ray scan technique.
Time Frame: DEXA scans were taken at Baseline (Day 1) and Week 48.
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy.
Measure: Mean (95% Confidence Interval); unit: grams/ centimeters ^2 (g/cm^2)
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 118 | 82
grams/ centimeters ^2 (g/cm^2)
  Bone Mineral Density of Both Arms | -1 [-1.9 to -0.4] | -1 [-2.1 to -0.4]
  Bone Mineral Density of Both Legs | -2 [-2.0 to -1.1] | -2 [-2.4 to -1.4]
  Bone Mineral Density of Trunk | -4 [-4.3 to -3.0] | -4 [-5.2 to -3.4]
  Bone Mineral Density of Total Body | -2 [-2.7 to -1.7] | -3 [-3.1 to -2.1]

64. Secondary Outcome: Mean Percent Changes From Baseline in BMD Measured by DEXA at Week 96
Description: as for outcome 63
Time Frame: Baseline (Day 1) and Week 96
Population: As-treated participants in the lipodystrophy substudy who participated in the substudy and signed the informed consent for the substudy.
Measure: Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 106 | 70
g/cm^2
  Bone Mineral Density of Both Arms | -1 [-2.3 to -0.5] | -2 [-3.2 to -1.2]
  Bone Mineral Density of Both Legs | -2 [-2.7 to -1.1] | -3 [-3.4 to -1.9]
  Bone Mineral Density of Trunk | -3 [-3.7 to -1.9] | -5 [-5.7 to -3.5]
  Bone Mineral Density of Total Body | -3 [-3.4 to -1.9] | -4 [-4.5 to -2.9]

65. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 96
Description: Mean change from baseline in weight at Week 96
Time Frame: Baseline (Day 1) and Week 96
Population: Safety analyses of the treatment period are based on treated population with values for this parameter.
Measure: Mean (Standard Error); unit: kg
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 361 | 338
kg | 5 (0.4) | 3 (0.3)

66. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 48
Description: Mean change from baseline in body weight at Week 48 was determined.
Time Frame: Baseline (Day 1) and Week 48
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy, and who had values for this parameter.
Measure: Mean (Standard Error); unit: kg
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 118 | 85
kg | 4 (0.5) | 3 (0.7)

67. Secondary Outcome: Mean Change From Baseline in BMI at Week 96
Time Frame: Baseline (Day 1) and Week 96
Population: Safety analyses of the treatment period are based on treated population with values for this parameter.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 359 | 338
kg/m^2 | 1.6 (0.13) | 1.0 (0.11)

68. Secondary Outcome: Mean Change From Baseline in Waist Circumference at Week 96
Description: Mean change From baseline in waist circumference at Week 96 was determined.
Time Frame: Baseline (Day 1) and Week 96.
Population: as for outcome 66
Measure: Mean (Standard Error); unit: cm
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 100 | 71
cm | 6 (0.8) | 2 (0.8)

69. Secondary Outcome: Mean Change From Baseline in Waist Circumference at Week 48
Description: Mean change from baseline in waist circumference at Week 48 was determined.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 66
Measure: Mean (Standard Error); unit: cm
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 109 | 77
cm | 4 (0.6) | 2 (0.7)

70. Secondary Outcome: Mean Change From Baseline in Waist-to-hip-ratio at Week 96
Description: Mean change from baseline in waist-to-hip-ratio at Week 96 was determined.
Time Frame: Baseline (Day 1) and Week 96
Population: as for outcome 66
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 71
ratio | 0.02 (0.006) | 0.01 (0.08)

71. Secondary Outcome: Mean Change From Baseline in BMI at Week 48
Description: Mean change from baseline in BMI at Week 48 was determined.
Time Frame: Baseline (Day 1) and Week 48.
Population: as for outcome 66
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 118 | 85
kg/m^2 | 1.5 (0.19) | 1.1 (0.23)

72. Secondary Outcome: Mean Change From Baseline in Waist-to-hip-ratio at Week 48
Description: Mean change from baseline in waist-to-hip-ratio at Week 48 was determined.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 66
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 108 | 77
ratio | 0.02 (0.008) | 0.01 (0.008)

73. Secondary Outcome: Percentage of Participants With Lipoatrophy at Week 96
Description: Lipoatrophy, redistribution of body fat was defined as >= 20% decrease in limb fat. The percentage of participants with lipoatrophy from baseline was determined.
Time Frame: Baseline (Day 1) and Week 96
Population: as for outcome 66
Measure: Number; unit: percentage of participants
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 106 | 70
percentage of participants | 5 | 7

74. Secondary Outcome: Mean Changes From Baseline in Body Weight at Week 96
Description: Mean change in body weight from baseline was determined.
Time Frame: Physical examination was performed at Baseline (Day 1) and Weeks 48 and 96.
Population: as for outcome 66
Measure: Mean (Standard Error); unit: kg
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 110 | 78
kg | 6 (0.7) | 3 (0.8)

75. Secondary Outcome: Mean Change From Baseline in BMI at Week 96
Description: Mean change From baseline in BMI at Week 96 was determined.
Time Frame: Baseline (Day 1) and Week 96
Population: As-treated participants in the lipodystrophy substudy who participated and signed the informed consent for the substudy, and with values for this parameter.
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 110 | 78
kg/m^2 | 2.0 (0.26) | 1.2 (0.28)

76. Primary Outcome: Mean Change From Baseline in Fasting Non-High Density Lipoprotein (HDL) Cholesterol Associated With RETN_097
Description: The change-from-baseline was defined as the difference between the averages of post-treatment time points (Weeks 48 and 96) and baseline. Association analysis for each SNP was performed using a minor allele carrier (MAC) composed of heterozygous and rare homozygous genotypes, and wild type (WT, common homozygous). False discovery rate (FDR)-adjusted (adj) p-values were calculated for each phenotype-genotype pair.
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: Participants with both genotypes and phenotypes available in the metabolic substudy. Phenotypes used in this analysis were from 3 time points: baseline (Week 0), Week 48, and Week 96. No additional multiple testing adjustment was applied for the number of phenotypes being analyzed.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
mg/dL
  Fasting Non-HDL Cholesterol: RETN_097 WT | 12.50 (2.82) | 26.98 (2.96)
  Fasting Non-HDL Cholesterol: RETN_097 MAC | 13.23 (5.56) | 52.28 (6.67)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting non-HDL cholesterol (phenotype) and the RETN_097 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_097 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.0847, linear mixed effect model — The explanatory variables in the model include treatment, genotype, time, and their interaction effects as fixed effects and the spatial exponential with respect to time from baseline was used to model the covariance structure of repeated measures; The FDR multiple testing adjustment was used to adjust p-values for the number of SNPs being tested (only SNPs with FDR-adj p-values <0.2 reported)

77. Primary Outcome: Mean Change From Baseline in Fasting Triglycerides Associated With RETN_097
Description: The change-from-baseline was defined as the difference between the averages of post-treatment time points (Weeks 48 and 96) and baseline. Association analysis for each SNP was performed using a minor allele carrier (MAC) composed of heterozygous and rare homozygous genotypes, and wild type (WT, common homozygous). False discovery rate (FDR)-adjusted p-values were calculated for each phenotype-genotype pair.
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
mg/dL
  Fasting Triglycerides: RETN_097 WT | 21.41 (8.6) | 68.06 (9.01)
  Fasting Triglycerides: RETN_097 MAC | 27.21 (16.9) | 157.87 (20.4)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting triglycerides (phenotype) and the RETN_097 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_097 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.0058, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

78. Primary Outcome: Mean Change From Baseline in Fasting Triglycerides Associated With RETN_2265
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
mg/dL
  Fasting Triglycerides: RETN_2265 WT | 19.61 (9.17) | 65.83 (9.36)
  Fasting Triglycerides: RETN_2265 MAC | 28.70 (14.5) | 148.95 (18.3)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting triglycerides (phenotype) and the RETN_2265 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, weeks 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_2265 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.0058, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

79. Primary Outcome: Mean Change From Baseline in Fasting Triglycerides Associated With RETN_598
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
mg/dL
  Fasting Triglycerides: RETN_598 WT | 20.23 (10.2) | 61.66 (10.5)
  Fasting Triglycerides: RETN_598 MAC | 25.78 (12.2) | 123.28 (14.2)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting triglycerides (phenotype) and the RETN_598 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_598 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.0253, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

80. Primary Outcome: Mean Change From Baseline in Fasting Triglycerides Associated With APOE_C130R
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
mg/dL
  Fasting Triglycerides: APOE_C130R WT | 23.27 (8.33) | 70.71 (9.52)
  Fasting Triglycerides: APOE_C130R MAC | 13.92 (26.0) | 131.56 (19.3)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting triglycerides (phenotype) and the APOE_C130R genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with APOE_C130R reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1173, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

81. Primary Outcome: Mean Change From Baseline in Fasting Triglycerides Associated With RETN_734
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
mg/dL
  Fasting Triglycerides: RETN_734 WT | 23.35 (8.67) | 75.12 (8.94)
  Fasting Triglycerides: RETN_734 MAC | 21.16 (20.4) | 155.28 (27.0)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting triglycerides (phenotype) and the RETN_734 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, weeks 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_734 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1173, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

82. Primary Outcome: Mean Change From Baseline in Fasting Plasminogen Activator Inhibitor (PAI)-1 Associated With APOE_R176C
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
ng/dL
  Fasting PAI-1: APOE_R176C WT | 5.98 (8.85) | 7.30 (9.90)
  Fasting PAI-1: APOE_R176C WT | -117.27 (37.3) | -5.94 (38.5)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting PAI-1 (phenotype) and the APOE_R176C genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, weeks 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with APOE_R176C reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1847, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

83. Primary Outcome: Mean Change From Baseline in Fasting Tumor Necrosis Factor (TNF)-Alpha Associated With IL6_5309
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
pg/mL
  Fasting TNF-alpha: IL6_5309 WT | -1.19 (2.24) | -2.68 (2.68)
  Fasting TNF-alpha: IL6_5309 MAC | 6.01 (1.47) | 1.41 (1.51)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis:There is no association between the mean change from baseline in fasting Tumor Necrosis Factor(TNF)-alpha (phenotype) and the IL6_5309 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, wk48 and 96) to test the overall genotype effect (ie. an omnibus test on both marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with IL6_5309 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1833, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

84. Primary Outcome: Mean Change From Baseline in Fasting Tumor Necrosis Factor (TNF)-Alpha Asssociated With RS11030679
Description: as for outcome 77
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
pg/mL
  Fasting TNF-alpha: RS11030679 WT | 7.58 (1.72) | -0.13 (1.73)
  Fasting TNF-alpha: RS11030679 MAC | 0.02 (1.72) | 1.27 (2.00)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in fasting TNF-alpha (phenotype) and the RS11030679 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_097 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1833, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

85. Primary Outcome: Mean Change From Baseline in Subcutaneous Adipose Tissue (SAT)-To-Trunk Adipose Tissue (TAT) Ratio Associated With CCDC122_5980
Description: The change-from-baseline was defined as the difference between the averages of post-treatment time points (Weeks 48 and 96) and baseline. Association analysis for each SNP was performed using a minor allele carrier (MAC) composed of heterozygous and rare homozygous genotypes, and wild type (WT, common homozygous). False discovery rate (FDR)-adjusted p-values were calculated for each phenotype-genotype pair. SAT and TAT were measured by computed tomography (CT).
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
cm^2
  SAT-to-TAT Ratio: CCDC122_5980 WT | 0.03 (0.01) | 0.03 (0.02)
  SAT-to-TAT Ratio: CCDC122_5980 MAC | 0.11 (0.02) | 0.02 (0.02)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in SAT-to-TAT Ratio (phenotype) and the CCDC122_5980 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with CCDC122_5980 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1694, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

86. Primary Outcome: Mean Change From Baseline in Visceral Adipose Tissue (VAT) Associated With BRUNOL_1842
Description: The change-from-baseline was defined as the difference between the averages of post-treatment time points (Weeks 48 and 96) and baseline. Association analysis for each SNP was performed using a minor allele carrier (MAC) composed of heterozygous and rare homozygous genotypes, and wild type (WT, common homozygous). False discovery rate (FDR)-adjusted p-values were calculated for each phenotype-genotype pair. VAT was measured by computed tomography (CT).
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
cm^2
  VAT: BRUNOL_1842 WT | 23.45 (6.55) | 10.38 (7.13)
  VAT: BRUNOL_1842 MAC | -3.20 (6.18) | -1.76 (9.32)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in VAT (phenotype) and the BRUNOL_1842 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, week 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with BRUNOL_1842 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1335, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

87. Primary Outcome: Mean Change From Baseline in VAT Associated With RETN_730
Description: as for outcome 86
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
cm^2
  VAT: RETN_730 WT | -2.95 (6.10) | 13.69 (8.03)
  VAT: RETN_730 MAC | 23.29 (6.52) | -1.05 (7.61)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in VAT (phenotype) and the RETN_730 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, weeks 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with RETN_730 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1335, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

88. Primary Outcome: Mean Change From Baseline in VAT-to-TAT Ratio Associated With CCDA122_5980
Description: The change-from-baseline was defined as the difference between the averages of post-treatment time points (Weeks 48 and 96) and baseline. Association analysis for each SNP was performed using a minor allele carrier (MAC) composed of heterozygous and rare homozygous genotypes, and wild type (WT, common homozygous). False discovery rate (FDR)-adjusted p-values were calculated for each phenotype-genotype pair. VAT and TAT were measured by computed tomography (CT).
Time Frame: Baseline (Day 1), Week 48, and Week 96.
Population: as for outcome 76
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD | LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD
Number analyzed (Participants) | 99 | 100
cm^2
  VAT-to-TAT Ratio: CCDA122_5980 WT | -0.03 (0.01) | -0.03 (0.02)
  VAT-to-TAT Ratio: CCDA122_5980 MAC | -0.11 (0.02) | -0.02 (0.02)
Statistical Analysis 1: Comparison: ATV 300 mg QD + RTV 100 mg QD + TDF 300 mg QD + FTC 200 mg QD vs LPV 400mg BID + RTV 100mg BID + TDF 300 mg QD + FTC 200 mg QD; Null Hypothesis: There is no association between the mean change from baseline in VAT-to-TAT Ratio (phenotype) and the CCDA122_5980 genotypes. A single SNP association analysis was conducted using the linear mixed effect model for repeated measures (baseline, weeks 48 and 96) to test the overall genotype effect (i.e. an omnibus test on both the marginal genotype effect and the genotype-by-treatment interaction effect). Number of participants with CCDA122_5980 reported in Outcome Measure 16; Test type: Superiority or Other; p = 0.1696, linear mixed effect model — [p-value comment as in outcome 76, analysis 1]; [statistical method as in outcome 76, analysis 1]

ADVERSE EVENTS:
Description: Number of SAEs presented here differs from those in Outcome Measures, as the treated population was used for this section, not the all enrolled population that was used for the Outcome Measures. The number of AEs presented here also differs from those in the Outcome Measure, as the AEs here do not include SAEs.
Groups:
- ATV/RTV/Tenofovir/Emtricitabine: Participants were administered an oral dose of Atazanavir (ATV) 300 mg and ritonavir (RTV) 100 mg once daily along with food. Doses were taken 24 hours apart at the same time as fixed dose combination tenofovir (TDF) 300 mg plus emtricitabine (FTC) 200 mg once daily.
- LPV/RTV/Tenofovir/Emtricitabine: Participants were administered lopinavir (LPV) 400 mg or ritonavir (RTV) 100 mg twice daily along with food. Doses were taken approximately 12 hours apart while tenofovir (TDF) 300 mg once daily and emtricitabine (FTC) 200 mg once daily was administered at the same time as 1 of the 2 daily doses of LPV/RTV.
Arm/Group | ATV/RTV/Tenofovir/Emtricitabine | LPV/RTV/Tenofovir/Emtricitabine
Serious Adverse Events (participants affected / at risk) | 61/441 | 48/437
Other Adverse Events (participants affected / at risk) | 355/441 | 370/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV/Tenofovir/Emtricitabine (N=441) | LPV/RTV/Tenofovir/Emtricitabine (N=437)
WEIGHT DECREASED (Investigations) | 1 | 3
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 1
ANXIETY (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 2 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLESTASIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 2 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
IMMUNE RECONSTITUTION SYNDROME (Immune system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 3 | 6
ENTERITIS (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
COLONIC STENOSIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1
MESENTERIC ARTERY THROMBOSIS (Gastrointestinal disorders) | 0 | 1
INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 3
SINUSITIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1
MENINGITIS (Infections and infestations) | 1 | 0
CANDIDIASIS (Infections and infestations) | 1 | 0
ORAL HERPES (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 2 | 0
TUBERCULOSIS (Infections and infestations) | 1 | 0
SALMONELLOSIS (Infections and infestations) | 0 | 1
TOXOPLASMOSIS (Infections and infestations) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 1
LOBAR PNEUMONIA (Infections and infestations) | 2 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
BULLOUS IMPETIGO (Infections and infestations) | 1 | 0
PERIANAL ABSCESS (Infections and infestations) | 0 | 1
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0
MENINGITIS BACTERIAL (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
CEREBRAL TOXOPLASMOSIS (Infections and infestations) | 1 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 3 | 2
MENINGITIS CRYPTOCOCCAL (Infections and infestations) | 2 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 | 1
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 | 1
PARASITIC GASTROENTERITIS (Infections and infestations) | 1 | 0
EXTRAPULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 1
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 1 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
MYCOBACTERIUM AVIUM COMPLEX INFECTION (Infections and infestations) | 1 | 2
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 3
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERLACTACIDAEMIA (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1
ADNEXA UTERI MASS (Reproductive system and breast disorders) | 1 | 0
FANCONI SYNDROME (Congenital, familial and genetic disorders) | 1 | 0
INJURY (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0
CHEST INJURY (Injury, poisoning and procedural complications) | 0 | 1
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ERGOT POISONING (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OEDEMA (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 3
ASTHENIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MEDULLOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
TESTICULAR NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN MALE REPRODUCTIVE TRACT NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV/RTV/Tenofovir/Emtricitabine (N=441) | LPV/RTV/Tenofovir/Emtricitabine (N=437)
OCULAR ICTERUS (Eye disorders) | 43 | 0
JAUNDICE (Hepatobiliary disorders) | 83 | 2
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 51 | 3
HEADACHE (Nervous system disorders) | 81 | 67
DIZZINESS (Nervous system disorders) | 34 | 29
NAUSEA (Gastrointestinal disorders) | 73 | 103
VOMITING (Gastrointestinal disorders) | 34 | 48
DIARRHOEA (Gastrointestinal disorders) | 108 | 236
DYSPEPSIA (Gastrointestinal disorders) | 24 | 27
ABDOMINAL PAIN (Gastrointestinal disorders) | 30 | 31
INFLUENZA (Infections and infestations) | 33 | 33
BRONCHITIS (Infections and infestations) | 37 | 29
PHARYNGITIS (Infections and infestations) | 17 | 23
HERPES ZOSTER (Infections and infestations) | 19 | 22
NASOPHARYNGITIS (Infections and infestations) | 66 | 73
URINARY TRACT INFECTION (Infections and infestations) | 24 | 22
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 37 | 54
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 19 | 48
RASH (Skin and subcutaneous tissue disorders) | 27 | 19
BACK PAIN (Musculoskeletal and connective tissue disorders) | 38 | 14
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 32 | 20
COUGH (Respiratory, thoracic and mediastinal disorders) | 28 | 34
PYREXIA (General disorders) | 25 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.